CLINICAL TRIAL: NCT07094490
Title: Comparison of Posture and Respiration in Adults With and Without Head Forward Posture
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, PhD, Nigde Omer Halisdemir University
Other Study IDs: E-86837521-050.99-579759
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FHP: participants with a craniocervical angle ≤ 50°
- control: participants with a craniocervical angle > 50°

SUMMARY:
Forward head posture (FHP) is defined as the position in which the head is in front of the shoulder and is one of the most common musculoskeletal problems caused by increasing computer and smartphone use. This study aims to compare spinal alignment, pulmonary function, and respiratory muscle strength between individuals with and without FHP.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-35

Exclusion Criteria:

* presence of diagnosed respiratory, neurological, orthopedic, psychiatric, or cardiac conditions; any limitations that could interfere with assessments; pregnancy or breastfeeding; a history of neck trauma; and previous surgery involving the neck or lower back

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with a CVA of 50 degrees and less than 50 degrees will be included in the head forward posture group, and participants with a CVA above 50 degrees will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Tests- FEV1/FVC | baseline
  The person will be asked to take a few normal breaths followed by as deep a breath as possible and instructed to exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FVC | baseline
  The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FEV1 | baseline
  The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- PEF | Baseline
  The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Respiratory Muscle Strength- MIP | Baseline
  For the MIP assessment, participants were instructed to perform a rapid and forceful inspiration following a maximal expiration. Each maneuver was sustained for at least 2-3 seconds.
Respiratory Muscle Strength- MEP | Baseline
  For MEP assessment, they were asked to exhale rapidly and forcefully following maximal inspiration. Each maneuver was sustained for at least 2-3 seconds.
Posture- Sagittal head angle | Baseline
  The Sagittal head angle is defined as the angle formed between a line passing through the canthus and the tragus and a horizontal line.
Posture-Craniovertebral angle | baseline
  Craniovertebral angle is defined as the angle formed by the intersection of a line connecting the spinous process of C7 to the tragus of the ear and a horizontal line.
Posture- Sagittal shoulder angle | Baseline
  Sagittal shoulder angle is the angle formed between a horizontal line passing through the midpoint of the humerus and a line connecting the midpoint of the humerus to the spinous process of C7
Posture- Kyphosis | Baseline
  Thoracic kyphosis angle was determined by measuring the angles between the spinous processes of the 1st-2nd Thoracic (T1-T2) vertebrae and the 12th Thoracic-1st Lumbar (T12-L1) vertebrae using the inclinometer.
Posture- Lordosis | Baseline
  Lumbar lordosis angle was determined by measuring the angles between the spinous processes of the T12-L1 and 2nd-3rd Sacral (S2-S3) vertebrae.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Demirtaş, PhD, Principal Investigator — Niğde Ömer Halisdemir Üniversitesi
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No